CLINICAL TRIAL: NCT05184270
Title: Integration of Auditory Slow-Wave Stimulation Into Subthalamic Deep Brain Stimulation to Enhance Deep Sleep in Parkinson's Disease: A Proof-of-Concept Study
Brief Title: Integration of Auditory, and Deep Brain Stimulation to Enhance Deep Sleep in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Baumann (Other)
Collaborators: Klinik Lengg, Zurich (Other); University Children's Hospital (Other); University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Christian Baumann, Professor, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PD-LFP-AS
Record Dates: First submitted 2021-10-15; First posted 2022-01-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: sleep; neurodegeneration; slow-wave sleep; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease; Nerve Degeneration | interventions — Acoustic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Measurements (Experimental): LFP recording from STN using externalized wires or implanted neurostimulator, while simultaneously recording clinical surface EEG and applying AS during deep sleep.
  Interventions: Device: Acoustic stimulation

INTERVENTIONS:
Device: Acoustic stimulation — In this project, the intervention is a presentation of low-volume non-arousing auditory stimuli during deep NREM sleep via attached headphones. Stimuli will be applied targeting the up-phase of slow waves to enhance sleep slow-wave activity.
  Previous studies showed that this procedure does not lead to reduced sleep quality nor result in changed sleep architecture. Therefore, no negative consequences as a result of our intervention are to be expected. In fact, it is currently applied in several other studies including children, adults, and the elderly. Importantly, stimulation is not arousing, as the sounds presented during deep sleep are brief (50 ms) and at low volume (around 50 dB). In case of arousal during sleep (detected using the surface EEG signal), the volume will be adjusted.

SUMMARY:
The study is an open-label trial to validate the local field potential (LFP) activity in the subthalamic nucleus (STN) for slow-wave detection during acoustic stimulation during nighttime sleep in Parkinson's disease patients that receive deep-brain-stimulation (DBS) therapy with the novel PERCEPT™ DBS system.

DETAILED DESCRIPTION:
The objective of this study is to validate the STN signal for slow-wave detection during auditory stimulation. To test this, the electrophysiological activity within the STN will be measured as local field potentials (LFP) using standard STN-DBS electrodes. To assess whether the recorded STN activity can be used for AS, the coherence analysis of cortical and STN slow waves will be performed.

At the screening consultation, the study physician will obtain written informed consent, confirm inclusion and exclusion criteria, and obtain entry questionnaires including demographics, medical history, and concomitant therapy. Following a successful screening consultation, the study physician will schedule a screening night at the sleep laboratory in the department of Neurology, University Hospital Zurich (USZ), during which clinical surface EEG (12-channel system, including EMG, ECG, and EOG) will be recorded and AS will be applied. To test the individual susceptibility to AS, ERPs to auditory stimuli and SWA change will be assessed.

If the screening night was successful, each patient will undergo a baseline consultation and 3 recording sessions.

During all 3 recording sessions, the patients will be asked about their subjective sleep quality and current mood, concomitant therapy (including LED), and MDS-UPDRS III will be performed by the study physician. The surgical implantation (which is not part of the current proposal) follows standardized clinical protocol and is applied in 2 steps. Sleep will be recorded simultaneously with clinical surface EEG and STN LFP in all 3 recording sessions (combined LFP-EEG recording) and AS will be performed based on slow-wave detected in the surface EEG.

In detail: In the first step, DBS leads are implanted in the STN, keeping the wires externalized. Following one night in the intensive or intermediate care unit for monitoring, patients will undergo a full-night combined LFP-EEG recording and AS (Recording Session 1), with LFP data collected from the externalized wires (DBS off). Next, the surgery will be completed by implantation of the neuromodulator and its connection to the DBS leads. Following the completion of the surgery, rehabilitation will start. The rehabilitation period will last for 2-5 weeks. At the end of the rehabilitation Recording Session 2 and 3 will take place. These recording session will be separated by 2-3 days and their order will be randomized and counterbalanced across participants. During Recording Session 2, combined LFP-EEG recording and AS will be performed during first 4 hours of the night sleep; STN LFP will be recorded with the implanted neurostimulator (DBS off). Recording Session 3 will be similar to Recording Session 2, but with DBS on (i.e. using DBS settings that were adjusted during rehabilitation). Because stable LFP recordings by PERCEPT™ PC neurostimulator is only possible for 4 hours, LFP sleep recordings during Recording Session 2 and 3 are limited to the first 4h of sleep. Surface EEG and AS, however, will be performed for the whole night after the LFP recoding end. Recording Sessions 2 and 3 will take place either at Clinic Lengg or in the USZ sleep laboratory (if the patient will be at a different rehabilitation center than Clinic Lengg).

Additionally, circadian rhythm will be assessed continuously throughout the interventions using actigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosis of PD along with international criteria with mild to moderate disease severity (Hoehn-Yahr (HY) stages ll-lll), selected for receiving STN-DBS therapy with the neurostimulator PERCEPT™
* Sufficient German language comprehension to follow the study procedures and answer all questions related to the study outcomes
* Age above 18 years
* Negative pregnancy test during screening in female patients of childbearing potential (except in women who are surgically sterilized/hysterectomized or post-menopausal for longer than 1 year)

Exclusion Criteria:

* Failure to give informed consent
* Known presence of neurologic (other than PD), psychiatric, or systemic diseases (others than associated with PD)
* Clinical moderate to severe sleep-wake disorders (e.g. RLS-Index≥20, sleep apnea index ≥ 15 or, PLM-Index ≥ 15 if associated with arousals assessed during clinical PSG (in the framework of the pre-DBS work-up) and the clinical presentation of a RLS)
* Atypical or secondary Parkinsonism
* Severe medical conditions as renal insufficiency, liver failure, or congestive heart failure
* Skin disorders/problems/allergies in face/ear area that could worsen with electrode application
* Regular use of benzodiazepines other long-acting central nervous system (CNS)-depressant substances or long-acting antidepressants
* Use of melatonin less than 1 day prior to recording session
* Substance or alcohol abuse (i.e. > 0.5 l wine or 1 l beer per day)
* High caffeine consumption (> 5 servings/day; including coffee, energy drink)
* Known or suspected drug- or medication abuse
* Hearing deficiency resulting in inability to hear the auditory stimuli during sleep (based on results of standard pure-tone threshold audiometry)
* Not tolerating AS during screening night
* Inability to follow the procedures of the study, e.g. due to language problems or cognitive deficits
* Participation in another study with the intervention within the 30 days preceding, and during the present study
* Previous enrolment in the current study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons
* Shift work (work during the night)
* Travelling more than 2 time zones in the last month before the intervention starts or during the intervention (start of intervention will be adapted to fit with this criteria)
* Lack of safe contraception, defined as: Female patients of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Please note that female patients who are surgically sterilized/hysterectomized or post-menopausal for longer than 1 year are not considered as being of child bearing potential.
* During DBS implantation/ICU:

  * Use of long-acting substances (i.e. long-lasting benzodiazepines, anti-depressants)
  * Use of full anesthesia
  * Atypical STN electrophysiology
  * Miss-location of the DBS leads (location will be checked after surgery using SureTune™ Medtronic software based on CT and MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Identification of STN LFP correlates of cortical slow waves (i.e. 1-4 Hz, in the surface EEG) | Through study completion, an average of 2 years
  The temporal relationships of the surface EEG and the LFP will be investigated using the event-related potentials (ERP) and cross-correlation analysis.
Comparing the slope of slow wave across the night between surface EEG and STN-LFP | Through study completion, an average of 2 years
  In the EEG and the LFP recordings slow waves (0.5-4.5Hz) will be detected during all night NREM sleep. The slope of all detected slow-waves at the beginning of the night (i.e., first hour of sleep) will be compared to the slope of all detected slow waves at the end of the night (i.e., last hour of sleep) for the EEG and the LFP recordings separately. The overnight difference will be compared between the EEG and the LFP recordings.
Comparing the amplitude of slow wave across the night between surface EEG and STN-LFP | Through study completion, an average of 2 years
  In the EEG and the LFP recordings slow waves (0.5-4.5Hz) will be detected during all night NREM sleep. The amplitude of all detected slow-waves at the beginning of the night (i.e., first hour of sleep) will be compared to the slope of all detected slow waves at the end of the night (i.e., last hour of sleep) for the EEG and the LFP recordings separately. The overnight difference will be compared between the EEG and the LFP recordings.
Comparing the incidence of slow wave across the night between surface EEG and STN-LFP | Through study completion, an average of 2 years
  In the EEG and the LFP recordings slow waves (0.5-4.5Hz) will be detected during all night NREM sleep. The number of all detected slow-waves at the beginning of the night (i.e., first hour of sleep) will be compared to the number of all detected slow waves at the end of the night (i.e., last hour of sleep) for the EEG and the LFP recordings separately. The overnight difference will be compared between the EEG and the LFP recordings.
AS effect on SWA in the surface EEG and STN-LFP | Through study completion, an average of 2 years
  Comparing SWA (EEG power between 0.5-4.5Hz) during ON and OFF windows between surface EEG and STN-LFP
AS effect on the slope of slow waves in the surface EEG and STN-LFP | Through study completion, an average of 2 years
  Comparing the slope of slow waves of all detected slow waves during ON compared to the slope of slow waves of all detected slow waves during OFF windows between surface EEG and STN-LFP
AS effect on the amplitude of slow waves in the surface EEG and STN-LFP | Through study completion, an average of 2 years
  Comparing the amplitude of slow waves of all detected slow waves during ON compared to the slope of slow waves of all detected slow waves during OFF windows between surface EEG and STN-LFP
AS effect on frequencies over >4Hz | Through study completion, an average of 2 years
  Comparing event-related potentials (ERP) between surface EEG and STN-LFP
AS effect on frequencies over >4Hz | Through study completion, an average of 2 years
  Comparing time-frequency analysis of event-related spectral power (ERSP) between surface EEG and STN-LFP
AS effect on frequencies over >4Hz | Through study completion, an average of 2 years
  Comparing inter-trial phase coherence (ITPC) between surface EEG and STN-LFP

SECONDARY OUTCOMES:
Quantitative comparison of presented stimuli between recording sessions (i.e. DBS ON vs DBS OFF), i.e., total number of stimuli presented | Through study completion, an average of 2 years
  Number of presented tones will be compared between Recording Session 1, 2 and 3
Quantitative comparison of presented stimuli between recording sessions (i.e. DBS ON vs DBS OFF), i.e., phase targeting of AS | Through study completion, an average of 2 years
  Accuracy of slow-wave phase targeting during AS will be compared between Recording Session 1, 2 and 3
Quantitative comparison of presented stimuli between recording sessions (i.e. DBS ON vs DBS OFF), i.e., characterization of detected slow-waves | Through study completion, an average of 2 years
  The slope of detected slow-waves will be compared between Recording Session 1,2 and 3
Quantitative comparison of presented stimuli between recording sessions (i.e. DBS ON vs DBS OFF), i.e., characterization of detected slow-waves | Through study completion, an average of 2 years
  the amplitude of detected slow-waves will be compared between Recording Session 1,2 and 3
Investigation of relationships between behavioral performance changes and the AS effects (slow-wave characteristics in surface EEG and STN LFP) under DBS ON and OFF conditions | Through study completion, an average of 2 years
  Comparing reaction time and response inhibition in the Go-NoGo Task between conditions and the evening and morning

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, University Hospital Zurich, Zurich, Switzerland